CLINICAL TRIAL: NCT05140980
Title: Sexuality Education: Knowledge of Women Aged 18 to 25
Acronym: EDUSEX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-006-EDUSEX
Record Dates: First submitted 2021-11-17; First posted 2021-12-02 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Sexual Behavior
Keywords: Sexuality; knowledge; young women; education
MeSH Terms: conditions — Sexual Behavior; Sexuality | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- "women aged 18 to 25" group: "women aged 18 to 25" group: women aged 18 to 25 with or without sexual activity
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — evaluation of women's knowledge concerning sexuality

SUMMARY:
Information, education and communication concerning sexual health are essential for enable to do informed and responsible decisions about it.

In France, education for sexuality in schools still remains unequal and is considered as unsuited to the realities of young people. This observation led to the development of a national sexual health strategy. One of the challenges is to promote and enhance the implementation of interdisciplinary sexuality education. Midwives are and should be involved in the issue of sexuality.

DETAILED DESCRIPTION:
The aim of the study is to describe knowledge concerning sexuality of young women aged 18 to 25.

ELIGIBILITY:
Inclusion Criteria:

* female
* aged 18 to 25 years old
* with or without sexual activity
* agreeing to participate in the study

Exclusion Criteria:

- none

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women aged 18 to 25
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Knowledge about clitoris | Day 0
  knowledge about the clitoris functions: reproduction (yes/no), sexual pleasure (yes/no), urinary finction (yes/no) and childbirth (yes/no)

SECONDARY OUTCOMES:
Sexual health well-being | Day 0
  Personal sexual fulfillment evaluated using a Likert scale (from "not at all" to "totally")

CONTACTS AND LOCATIONS:
Locations (1):
- Cabinet de Sage Femme Liberale, Reims, Grand Est, France